CLINICAL TRIAL: NCT01951417
Title: Epiduo® (Adapalene and Benzoyl Peroxide) Gel 0.1%/2.5% Pump Cetaphil® DermaControl™ Moisturizer SPF 30, and Cetaphil® DermaControl™ Foaming Wash Regimen in Patients With Mild to Moderate Acne Vulgaris
Brief Title: Adapalene BPO Gel Pump, Moisturizer SPF 30 and Foam Wash in Patients With Mild to Moderate Acne Vulgaris
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: GLI.04.SRE.04.US10268
Record Dates: First submitted 2013-09-23; First posted 2013-09-26 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2022-08-23 (Actual); Status verified 2016-02

CONDITIONS: Acne
MeSH Terms: conditions — Acne Vulgaris | interventions — Adapalene, Benzoyl Peroxide Drug Combination; Adapalene; Benzoyl Peroxide; Gels

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adapalene/BPO Gel/Foam Wash/Moisturizer (Experimental): Adapalene BPO Gel Pump (once daily) in conjunction with a Foam Wash (twice daily) and Moisturizer SPF 30 (once daily)
  Interventions: Drug: Adapalene/BPO Gel; Other: Moisturizer SPF 30; Other: Foam Wash

INTERVENTIONS:
Drug: Adapalene/BPO Gel — Adapalene/Benzoyl Peroxide (BPO) Gel Pump (once daily)
  Other Names: Epiduo® (adapalene and benzoyl peroxide) Gel 0.1%/2.5% Pump; Adapalene and benzoyl peroxide (BPO) gel
Other: Moisturizer SPF 30 — Moisturizer SPF 30 (once daily)
  Other Names: Cetaphil® DermaControl™ Moisturizer SPF 30
Other: Foam Wash — Foam Wash (twice daily)
  Other Names: Cetaphil® DermaControl™ Foam Wash

SUMMARY:
This is an open-label, multi-center study to be conducted in the United States. The study will examine the change in lesion count in subjects using Epiduo® Gel Pump (once daily) in conjunction with Cetaphil® DermaControl™ Foam Wash (twice daily) and Moisturizer SPF 30 (once daily). Subjects with a clinical diagnosis of mild or moderate acne who are eligible for treatment with Epiduo® in accordance with the currently approved product labeling and who meet other inclusion/exclusion criteria are to be enrolled in the study and receive the study products for 8 weeks. Efficacy and safety assessments include: complete lesion counts, cutaneous irritation assessment, end of study treatment questionnaire, photographic evaluation for oiliness, skin tone, and P Acnes, hydration assessment, barrier function assessment, treatment compliance, and adverse event assessment.

ELIGIBILITY:
Inclusion Criteria:

- Men and women of any race, 9 years or older, with a diagnosis of mild to moderate acne, who are eligible for treatment with adapalene BPO gel in accordance with the currently approved product labeling.

Exclusion Criteria:

- Subjects with nodules and cysts, pregnant or breastfeeding, with any systemic or dermatological disorder, or topical condition or facial hair that could interfere with evaluations.

Min Age: 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2013-10; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua M Berlin, MD, Principal Investigator — Dermatology Associates, PA, of the Palm Beaches
Locations (5):
- United States (5):
  - Study Protocol, Inc., Boynton Beach, Florida
  - Tennessee Clinical Research Center, Nashville, Tennessee
  - Stephens & Associates, Carrollton, Texas
  - J&S Studies, Inc., College Station, Texas
  - The Dermatology Clinical Research Center of San Antonio, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Started | 81
Completed | 72
Not Completed | 9
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 6

BASELINE CHARACTERISTICS:
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Number analyzed (Participants) | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.0 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Safety Population
  Participants
    Female | 40
    Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 24
  White | 48
  More than one race | 0
  Unknown or Not Reported | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17
  Not Hispanic or Latino | 64
  Unknown or Not Reported | 0
Skin Type [Number; unit: participants]
  Dry | 5
  Normal | 22
  Oily | 32
  Combination | 22
Fitzpatrick Skin Type [Number; unit: participants] — Investigator assessment based on the standard Fitzpatrick Skin Type Scale (I to VI).
  TYPE 1: Highly sensitive, always burns, never tans. TYP E 2: Very sun sensitive, burns easily, tans minimally. TYPE 3: Sun sensitive skin, sometimes burns, slowly tans to light brown. TYPE 4: Minimally sun sensitive, burns minimally, always tans to moderate brown.
  TYPE 5: Sun insensitive skin, rarely burns, tans well. TYPE 6: Sun insensitive, never burns, deeply pigmented.
  --------------------------------------------------------------------------------
  participants
    I | 3
    II | 20
    III | 16
    IV | 19
    V | 13
    VI | 10
History of Acne [Mean (Standard Deviation); unit: years] | 4.4 (4.7)

OUTCOME MEASURES:

1. Primary Outcome: Total Lesion Count
Description: The change in total lesion count after use of adapalene BPO gel in conjunction with Foam Wash and Moisturizer SPF 30 for 2 weeks, 4 weeks, and 8 weeks.
Time Frame: Baseline, 2, 4, and 8 weeks
Population: ITT population (all subjects who had at least 1 post-treatment administration evaluation)
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Number analyzed (Participants) | 77
lesions
  Baseline | 76.7 (21.1)
  Week 2 | 53.9 (25.5)
  Week 4 | 50.0 (27.8)
  Week 8 | 43.7 (22.7)

2. Secondary Outcome: Inflammatory Lesions
Description: The change in inflammatory lesions after use of adapalene BPO gel in conjunction with Foam Wash and Moisturizer SPF 30 for 2 weeks, 4 weeks, and 8 weeks.
Time Frame: Baseline, 2, 4, and 8 weeks
Population: ITT population (all subjects who had at least 1 post-treatment administration evaluation)
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Number analyzed (Participants) | 77
lesions
  Baseline | 27.3 (6.4)
  Week 2 | 17.4 (9.0)
  Week 4 | 15.7 (11.3)
  Week 8 | 14.4 (9.5)

3. Secondary Outcome: Non-inflammatory Lesions
Description: The change in non-inflammatory lesions after use of adapalene BPO gel in conjunction with Foam Wash and Moisturizer SPF 30 for 2 weeks, 4 weeks, and 8 weeks
Time Frame: Baseline, 2, 4, and 8 weeks
Population: ITT population (all subjects who had at least 1 post-treatment administration evaluation)
Measure: Mean (Standard Deviation); unit: lesions
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Number analyzed (Participants) | 77
lesions
  Baseline | 49.4 (18.3)
  Week 2 | 36.4 (21.5)
  Week 4 | 34.1 (23.4)
  Week 8 | 29.2 (18.3)

4. Secondary Outcome: Subject Questionnaire
Description: Describe subject satisfaction after use of adapalene BPO gel in conjunction with Foam Wash and Moisturizer SPF 30 for 8 weeks.
Time Frame: Baseline, 2, 4, and 8 weeks
Population: ITT population (all subjects who had at least 1 post-treatment administration evaluation)
Measure: Number; unit: participants
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Number analyzed (Participants) | 77
participants
  Very satisfied | 23
  Satisfied | 42
  Undecided | 5
  Dissatisfied | 3
  Very dissatisfied | 1
  Missing | 3

5. Other Pre Specified Outcome: Erythema
Description: Cutaneous irritability assessments (stinging/burning, erythema, scaling, dryness) experienced during use of adapalene BPO gel in conjunction with Foam Wash and Moisturizer SPF 30 for 8 weeks.
Time Frame: Baseline, 2, 4, and 8 weeks
Population: As observed population
Measure: Number; unit: participants
Groups:
- Baseline; Week 2; Week 4; Week 8: Adapalene BPO Gel Pump (once daily) in conjunction with a Foam Wash (twice daily) and Moisturizer SPF 30 (once daily)
  * Adapalene/BPO Gel: Adapalene/Benzoyl Peroxide (BPO) Gel Pump (once daily)
  * Moisturizer SPF 30: Moisturizer SPF 30 (once daily)
  * Foam Wash: Foam Wash (twice daily)
Arm/Group | Baseline | Week 2 | Week 4 | Week 8
Number analyzed (Participants) | 81 | 76 | 76 | 72
participants
  None | 50 | 49 | 45 | 52
  Mild | 28 | 20 | 26 | 18
  Moderate | 3 | 7 | 5 | 2
  Severe | 0 | 0 | 0 | 0

6. Other Pre Specified Outcome: Scaling
Description: as for outcome 5
Time Frame: Baseline, 2, 4, and 8 weeks
Population: As observed population
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8
Number analyzed (Participants) | 81 | 76 | 76 | 72
participants
  None | 73 | 57 | 65 | 63
  Mild | 8 | 15 | 9 | 9
  Moderate | 0 | 4 | 2 | 0
  Severe | 0 | 0 | 0 | 0

7. Other Pre Specified Outcome: Dryness
Description: as for outcome 5
Time Frame: Baseline, 2, 4, and 8 weeks
Population: As observed population
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8
Number analyzed (Participants) | 81 | 76 | 76 | 72
participants
  None | 71 | 45 | 56 | 60
  Mild | 10 | 22 | 19 | 11
  Moderate | 0 | 9 | 1 | 1
  Severe | 0 | 0 | 0 | 0

8. Other Pre Specified Outcome: Stinging/Burning
Description: as for outcome 5
Time Frame: Baseline, 2, 4, and 8 weeks
Population: As observed population
Measure: Number; unit: participants
Arm/Group | Baseline | Week 2 | Week 4 | Week 8
Number analyzed (Participants) | 81 | 76 | 76 | 72
participants
  None | 80 | 48 | 63 | 62
  Mild | 1 | 23 | 12 | 10
  Moderate | 0 | 5 | 1 | 0
  Severe | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Adapalene/BPO Gel/Foam Wash/Moisturizer
Serious Adverse Events (participants affected / at risk) | 0/81
Other Adverse Events (participants affected / at risk) | 13/81
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adapalene/BPO Gel/Foam Wash/Moisturizer (N=81)
Erythema (Skin and subcutaneous tissue disorders) | 6 (6)
Dry skin (Skin and subcutaneous tissue disorders) | 4 (4)
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Skin burning sensatation (Skin and subcutaneous tissue disorders) | 1 (1)
Pain (General disorders) | 2 (2)
Muscle strain (Injury, poisoning and procedural complications) | 1 (1)
Accidental exposure to product by child (Injury, poisoning and procedural complications) | 1 (1)

LIMITATIONS AND CAVEATS:
* Open label study with small sample size
* Short study duration

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less